CLINICAL TRIAL: NCT03802084
Title: A Phase 1b/2a, Open-label, Multicentre Study to Assess the Safety, Tolerability, Pharmacokinetics, and Antitumor Activity of Vactosertib in Combination With Imatinib in Patients With Advanced Desmoid Tumor (Aggressive Fibromatosis)
Brief Title: A Study to Evaluate the Safety and Efficacy of Vactosertib and Imatinib in Patients With Advanced Desmoid Tumor
Status: Completed | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Hyo Song Kim (Other)
Responsible Party: Sponsor-Investigator, Hyo Song Kim, professor, Yonsei University
Organization: Yonsei University (Other)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 4-2018-0807
Record Dates: First submitted 2019-01-07; First posted 2019-01-14 (Actual); Last update posted 2024-05-13 (Actual); Status verified 2024-05

CONDITIONS: Desmoid Tumor
MeSH Terms: conditions — Desmoid Tumors | interventions — vactosertib

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- vactosertib/imatinib combination (Experimental)
  Interventions: Drug: vactosertib/imatinib combination

INTERVENTIONS:
Drug: vactosertib/imatinib combination — Phase 1 : Imatinib 400mg QD P q28days Vactosertib 1 cohort 200mg bid (D1-5, 8-12, 15-19, 22-26)
  * 1 cohort 100mg bid Phase 2 : Imatinib 400mg QD PO q28days. Vactosertib RP2D, bid (D1-5, 8-12, 15-19, 22-26)

SUMMARY:
This is a phase I/II, open-label, non-randomized, multicentre study to evaluate the clinical activity of vactosertib plus imatinib in desmoid tumor. Based on the background, TGF-β inhibition as a potential therapeutic target for desmoid tumor and convey significant implications for the clinical development. Therefore, investigator will conduct the phase II trial of vactosertib in combined with imatinib in desmoid tumor.

DETAILED DESCRIPTION:
Desmoid tumor (aggressive fibromatosis) is a mesenchymal neoplasm associated with mutations, resulting in -catenin-mediated transcriptional activation. It is composed of a clonal proliferation of mesenchymal, fibroblast-like cells occurred sporadic or as a part of familial adenomatosis polyposis. This tumor has high local recurrence rate after complete excision (~40%). Therefore, although lacking metastatic capability, patients experience repeated recurrence with attendant severe morbidity. Various systemic therapy using NSAID, cytotoxic agent (doxorubicin and vinblastine), biologic agents (tamoxifen, low-dose interferon), and tyrosine kinase inhibitors (imatinib) are recommended with modest activity. Among them, imatinib has shown promising activity and approved as standard treatment for desmoid tumor. However, still there is modest response (10-15% responses) and further combination strategy is warranted to improve antitumor efficacy.

The transforming growth factor-β (TGF-β) family of cytokines has 33 members in humans, including TGF-β isoforms, activins, bone morphogenetic proteins (BMPs), and growth and differentiation factors (GDFs). These factors regulate growth, survival, differentiation and migration of cells, and have important roles during embryonal development and in the control of adult tissue homeostasis. During carcinogenesis, TGF-β has a dual role; initially it suppresses tumorigenesis by inducing growth arrest and promoting apoptosis, however, in advanced cancers, where TGF-β often is overexpressed. In addition, TCGA (the cancer genome atlas) pan-cancer also demonstrated high expression of TGF-β responsive signature in desmoid tumor. Regarding the combination, TEW-7197 (vactosertib), a TGF-β inhibitor and imatinib demonstrated synergistic effect in vitro and xenograft model. Compared to imatinib alone, administration of imatinib plus vactosertib to mice significantly delayed disease relapse and prolonged survival. Collectively, these results indicate that vactosertib may be a promising candidate for a new therapeutic strategy.

Based on the background, TGF-β inhibition as a potential therapeutic target for desmoid tumor and convey significant implications for the clinical development. Therefore, investigator will conduct the phase II trial of vactosertib in combined with imatinib in desmoid tumor.

ELIGIBILITY:
Inclusion Criteria:

1. Histologically confirmed desmoid tumor (aggressive fibromatosis) not available for local treatment (surgical resection or radiation therapy)
2. Eastern Cooperative Oncology Group performance status of 0-1
3. Measurable lesion (RECIST 1.1.)
4. Patients with sufficient organ function according to laboratory findings

   * Hemoglobin ≥ 9.0 g/dL
   * Neutrophils ≥ 1000 /µL
   * Platelets ≥ 75,000/µL
   * Total Bilirubin ≤ 1.5 × UNL (upper normal limit): For patients with liver metastases, ≤2
   * Serum creatinine ≤1.5 X ULN or > 1.5 X Creatinine Clearance ≥50 mL/min for ULN patients (based on 24-hour urinalysis or Cockroft-Gault Formula calculations)
   * AST(SGOT)/ALT(SGPT) ≤ 3.0 × UNL or ≤ 5.0 × UNL (for patients with liver or bone metastases)
   * Alkaline Phosphatase (ALP): ≤ 3.0 × UNL or ≤ 5.0 × UNL (for patients with liver or bone metastases)
5. All patients must be able to provide a newly acquired tumor biopsy during screening (preferred) or provide an available tumor sample taken ≤3 years prior to screening.
6. Subjects must have ejection fraction ≥ 50% and no clinically significant valvular dysfunction

Exclusion Criteria:

1. Previous TGF-β inhibitor exposed patient
2. Patient who has had chemotherapy, radiotherapy, or biological therapy within 2 weeks
3. Any unresolved chronic toxicity greater than grade 2 from previous anticancer therapy.
4. Has an active infection requiring systemic therapy
5. Uncontrolled intercurrent illness, including symptomatic congestive heart failure (NYHA Class III/IV), uncontrolled hypertension (≥150/90mmHg), unstable angina pectoris or myocardial infarction (≤ 6 months prior to screening), uncontrolled cardiac arrhythmia, cardiac valulopathy
6. Uncontrolled or active central nervous system metastasis and/or carcinomatous meningitis
7. Child-Pugh B or C liver cirrhosis
8. History of another primary malignancy.
9. Female patients who are pregnant or breastfeeding or male or female patients of reproductive potential who are not willing to employ effective birth control from screening to 90 days after the last dose of investigational product(IP).
10. Major surgical procedure (as defined by the Investigator) within 28 days prior to the first dose of investigational product(IP).
11. Current or prior use of immunosuppressive medication within 14 days before the first investigational product(IP).

Min Age: 19 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 24 (Actual)
Dates: Start 2019-04-15 (Actual); Primary Completion 2024-03-26 (Actual); Study Completion 2024-03-26 (Actual)

PRIMARY OUTCOMES:
adverse event | 4 weeks
  to evaluate the safety and tolerability
clinical benefit rate was determined using RECIST 1.1 | 16weeks
  to evaluate antitumor activity by determining progression-free survival

CONTACTS AND LOCATIONS:
Locations (1):
- Severance Hospital, Yonsei University Health System, Seoul, South Korea

IPD SHARING:
Plan to Share IPD: No